CLINICAL TRIAL: NCT05863364
Title: Rifaximin for Preventing Progression and Complications in Patients With Decompensated Liver Cirrhosis: a Multi-center Randomized Prospective Study
Brief Title: Rifaximin for Preventing Progression and Complications in Patients With Decompensated Liver Cirrhosis
Acronym: RPPCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xin Zeng (Other)
Responsible Party: Sponsor-Investigator, Xin Zeng, Director of the department of gastroenterology, Shanghai East Hospital
Organization: Shanghai East Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DFYY2022096
Record Dates: First submitted 2022-12-28; First posted 2023-05-18 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-05

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Group A: Patients in the control group were administered only conventional therapy
- the low-dose rifaximin treatment group (Experimental): Group B
  Interventions: Drug: Low-dose of Rifaximin
- the conventional dose rifaximin treatment group (Experimental): Group C
  Interventions: Drug: Conventional dose of Rifaximin

INTERVENTIONS:
Drug: Low-dose of Rifaximin — The patients in group B were given rifaximin with the dose of 600mg/d (600mg, qd) for 24 weeks
  Other Names: Low-dose of Xifaxan
  Arms: the low-dose rifaximin treatment group
Drug: Conventional dose of Rifaximin — the patients in group C were delivered 1200mg/d (600mg, bid) for 24 weeks
  Other Names: Conventional dose of Xifaxan
  Arms: the conventional dose rifaximin treatment group

SUMMARY:
It is still not clear whether rifaximin can prevent the progression of liver cirrhosis, reduce the overall complications and improve the survival in patients with decompensated cirrhosis. This is a multi-center open-labelled randomized prospective study to evaluate the efficacy and safety of rifaximin in preventing the progression and complications in cirrhotic patients, and explore its reasonable dosage and possible mechanism. A total of 150 patients with decompensated liver cirrhosis will be enrolled in the study and randomly divided into three groups (the control group (A), the low-dose rifaximin treatment group (B), and conventional dose rifaximin treatment group (C)) with a ratio of 1:2:2. The patients in group B are given rifaximin with the dose of 600mg/d (600mg, qd) for 24 weeks, and the patients in group C are delivered 1200mg/d (600mg, bid) of rifaximin .During the entire study period, all other therapeutic strategies are kept unchanged in all the groups as long as possible. The proportion of patients with progression of cirrhosis, the incidence of total complications and each complication, survival rate and time, liver function and adverse events will be compared among the three groups. This study might provide a new feasible method with clinical application prospects for preventing the progression and reducing the incidence of liver cirrhosis related complications, improve the prognosis of patients with decompensated liver cirrhosis, and save medical resources.

DETAILED DESCRIPTION:
Rifaximin has been recommended as a prophylactic drug for hepatic encephalopathy (HE) and spontaneous bacterial peritonitis (SBP), the two major complications of liver cirrhosis. However, it is still not clear whether rifaximin can prevent the progression of liver cirrhosis, reduce the overall complications and improve the survival in patients with decompensated cirrhosis. Additionally, the role of rifaximin in the treatment of liver cirrhosis has not been fully clarified. We designed a multi-center open-labelled randomized prospective study to evaluate the efficacy and safety of rifaximin in preventing the progression and complications in cirrhotic patients, and explore its reasonable dosage and possible mechanism. A total of 150 patients with decompensated liver cirrhosis will be enrolled in the study. They will be randomly divided into three groups (the control group (A), the low-dose rifaximin treatment group (B), and conventional dose rifaximin treatment group (C)) with a ratio of 1:2:2. The patients in group B are given rifaximin with the dose of 600mg/d (600mg, qd) for 24 weeks, and the patients in group C are delivered 1200mg/d (600mg, bid) of rifaximin .During the entire study period, all other therapeutic strategies, such as antiviral agents, non-selective beta-blockers, liver protectants, and diuretics, are kept unchanged in all the groups as long as possible. The proportion of patients with progression of cirrhosis, acute decompensation, acute-on-chronic liver failure (ACLF), decompensation and stable decompensated cirrhosis, the incidence of total complications and each complication, survival rate and time, liver function and adverse events will be compared among the three groups. This study might provide a new feasible method with clinical application prospects for preventing the progression and reducing the incidence of liver cirrhosis related complications, improve the prognosis of patients with decompensated liver cirrhosis, and save medical resources.

ELIGIBILITY:
Inclusion Criteria:

* With a clinical diagnosis of decompensated liver cirrhosis on the basis of typical clinical manifestations, laboratory tests, imaging appearances and/or representative pathology results of liver biopsy. Decompensation of the disease was defined by at least having an episode of severe complications, including ascites, SBP, EGVB and HE.

Exclusion Criteria:

* Episodes of overt HE, EGVB or SBP within 4 weeks before the screening visit
* Uncontrolled severe infection or antibiotic use within 2 weeks before the screening visit
* Hepatitis B virus (HBV) DNA ≥ 500 copy/mL，or receipt of standard antiviral treatment for hepatitis B for less than 12 months
* Receiving antiviral treatment for hepatitis C or receipt of antiviral treatment for hepatitis C within 12 months before the screening visit
* If patients with autoimmune liver disease have been treated with ursodeoxycholic acid, hormone or other immunosuppressants, the dose stability time is less than 6 months
* With history of alcoholism in the last 12 weeks or unwilling to stop alcohol abuse after inclusion (≥ 20 g/day for women or ≥ 30 g/day for men)
* With confirmed or suspected malignancies
* Severe jaundice (serum total bilirubin level ≥ 85 μmol/L)
* Obvious renal dysfunction (serum creatinine ≥ 1.2-fold of upper normal limits)
* Severe electrolyte abnormality (serum sodium level < 125 mmol/L )
* Life-threatening leucocytopenia (white blood cell count < 1 × 10^9/L )
* Poorly controlled hypertension, diabetes mellitus or other severe heart and respiratory diseases (NYHA Ⅲ/Ⅳ, COPD GOLD C)
* With drug abuse, methadone treatment, drug dependence or mental illness
* HIV seropositivity
* Known to be allergic to rifaximin
* Pregnant and lactating women or women who do not rule out pregnancy
* Those who have participated in other drug trials within 12 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-18 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with progression of liver cirrhosis | 24 weeks
  The proportion of patients with progression of liver cirrhosis, which is defined as at least one additional stage of liver cirrhosis staging during the 24-week treatment phase

SECONDARY OUTCOMES:
Incidence of overall complications resulting from decompensated liver cirrhosis | 12 and 24weeks
  The incidence of overall complications resulting from decompensated liver cirrhosis in 12weeks and 24weeks, including refractory ascites, SBP, esophageal and gastric variceal bleeding (EGVB), overt hepatic encephalopathy(OHE), cute renal injury (AKI)/hepatorenal syndrome (HRS), primary hepatic carcinoma (PHC), etc.
Incidence of various complications of liver cirrhosis, including: refractory ascites, SBP, EGVB, OHE, AKI/HRS, PHC, etc. | 12 weeks and 24 weeks
  The incidence of each complication resulting from decompensated liver cirrhosis in 12weeks and 24weeks, including refractory ascites, SBP, EGVB, OHE, AKI/HRS, PHC, etc.
The proportion of patients with progression of liver cirrhosis | 12 weeks
  The proportion of patients with progression of liver cirrhosis, which is defined as at least one additional stage of liver cirrhosis staging during the 12-week treatment phase
The proportion of patients with acute decompensated (AD) | 12 and 24 weeks
  The proportion of patients with acute decompensated (AD)
The proportion of patients with stable decompensated cirrhosis | 24 weeks
  The proportion of patients with stable decompensated cirrhosis, which is defined as patients with decompensated cirrhosis who, while receiving sustained prophylaxis with diuretics, and/or lactulose or rifaximin, and/or non-selective beta-blockers or repeated endoscopic treatment of esophagogastric varices, do not present episodes of AD for a long-time period.
The proportion of patients with recompensation of cirrhosis | 24 weeks
  The proportion of patients with recompensation of cirrhosis, which is defined as the clinical phase of the disease prior to the resolution of cirrhosis induced by successful treatment of the underlying aetiology.
All-cause mortality | 24 weeks
  All-cause mortality during the 24-week treatment phase
Complication-free survival time | 24 weeks
  Complication-free survival time during the treatment phase
Liver transplantation free survival time | 24 weeks
  Liver transplantation free survival time during the treatment phase
Child-Pugh score | 24 weeks
  Liver function reflected by Child-Pugh score. A higher Child-Pugh score mean a worse outcome
The proportion of patients with different Child-Pugh class | 24 weeks
  The proportion of patients with Child-Pugh A/B/C （Child-Pugh A: Child-Pugh score<7; Child-Pugh B: Child-Pugh score 7~9; Child-Pugh C: Child-Pugh score>9 ）
Model for end-stage liver disease (MELD) score | 24 weeks
  Liver function reflected by MELD score. A higher MELD score mean a worse outcome

OTHER OUTCOMES:
Incidence of ACLF | 24 weeks
  The proportion of patients with ACLF during the treatment phase
Health-related quality of life (HRQoL) | 24 weeks
  HRQoL evaluated with chronic liver disease questionnaire,CLDQ)
Sarcopenia | 24 weeks
  Sarcopenia evaluated with L3 skeletal muscle index (L3-SMI) based on CT or MRI
Myosteatosis | 24 weeks
  Myosteatosis evaluated with L3 skeletal muscle density (L3-SMD) based on CT or MRI

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zeng, Dr., Principal Investigator — Department of Gastroenterology, Shanghai East Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No